CLINICAL TRIAL: NCT04685720
Title: A Pilot Study to Assess the Effect of Intermittent Inhaled Nitric Oxide on the Treatment of Nontuberculous Mycobacteria (NTM) Lung Infection in Cystic Fibrosis and Non-Cystic Fibrosis Patients
Brief Title: A Pilot Study to Assess the Effect of Intermittent iNO on the Treatment of NTM Lung Infection in CF and Non-CF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA_NTM_AU_01.01
Record Dates: First submitted 2020-12-07; First posted 2020-12-28 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia; Cystic Fibrosis; Mycobacterial Pneumonia; Mycobacterium Abscessus Infection; Mycobacterium Avium Complex
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous; Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled NO delivered using LungFit (Experimental): Inhaled Nitric Oxide in doses up to 250 ppm
  Interventions: Device: LungFit

INTERVENTIONS:
Device: LungFit — LungFit for NTM is an experimental device that produces Nitric Oxide from the ambient air.

SUMMARY:
The purpose of this open-label, multicenter, non-randomized, pilot study is to assess the safety of high dose intermittent iNO for treatment of NTM infection in CF and non-CF patients.

DETAILED DESCRIPTION:
The study will include 20 patients from up to four clinical sites in Australia. The overall treatment plan includes 2 weeks of inhalation treatments (intensive phase) of iNO four times per day at 4.5-hour intervals followed by 10 weeks of inhalation treatments (maintenance phase) at the maximum tolerated dose (a maximum of 250 ppm NO) inhaled twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with refractory NTM (MAC or MAbs) pulmonary infection
* CF and Non-CF patients

Exclusion Criteria:

* Diagnosis of methemoglobinemia or MetHb ≥2% at screening; treatment with any drug known to increase MetHb; known or suspected hemoglobinopathy.
* History of or current myeloproliferative disease, leukemia or other hematological malignancy; known or suspected immunodeficiency disease.
* Subjects with advanced cardiovascular disease or CHF
* Use of an investigational drug during the 30 days prior to enrollment.
* History of frequent epistaxis (>1 episode/month); significant hemoptysis (during the 30 days prior to enrollment.
* Subject on non-constant dose of systemic steroids within 30 days prior to enrollment; subjects on constant systemic steroids if the daily dose is higher than 10 mg/d prednisolone or equivalent.
* Active pulmonary malignancy (primary or metastatic) or any malignancy; history of lung transplantation.
* Pulmonary tuberculosis requiring treatment or treated within 2 years prior to screening.
* Uncontrolled hypertension within 3 months prior to or at screening
* Diagnosis of significant pulmonary hypertension indicated on echocardiogram at screening
* Clinically significant renal or liver laboratory abnormalities
* History of daily, continuous oxygen supplementation.
* Women of childbearing potential - pregnant or breastfeeding, or not on medically acceptable double methods of contraception from enrollment until Day 84.
* Smoking tobacco or any substance within 6 months prior to screening or anticipated inability to refrain from smoking throughout the study.
* Patient receiving drugs that have a contraindication with NO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent SAEs | Day 1 to Day 84
  The primary endpoint of the study is the number of patients with treatment-emergent SAEs

SECONDARY OUTCOMES:
Changes in NTM bacterial load from baseline to Day 174 | Day 1 to Day 174
  Changes in NTM bacterial load will be assessed by sputum culture in liquid and solid media.
Number of patients with culture conversion at Day 174 | Day 1 to Day 174
  NTM culture conversion will be defined as having at least three consecutive negative NTM cultures
Changes in quality of life assessed by CFQ-R for or QOL-B with NTM module | Day 1 to Day 174
  Changes in quality of life assessed by Cystic Fibrosis Questionnaire Revised [CFQ R] for CF patients or Quality of Life Questionnaire-Bronchiectasis [QOL-B] with NTM module for non-CF patients.
Changes in FEV1 from baseline to Day 174 | Day 1 to Day 174
  Respiratory function will be assessed by spirometry including FEV1.
Changes in activity tracker data as assessed by changes in distance from baseline to Day 174. | Day 1 to Day 174
  Patients will collect activity tracker data from 2 weeks before treatment and from Day 1 to Day 174.
Change in 6 Minute Walking Test | Day 1 to Day 84
  Change in 6 Minute Walking Test will be assessed by changes in distance between baseline and Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Gallipoli Medical Research Foundation, Greenslopes, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No